CLINICAL TRIAL: NCT04226443
Title: The Use of Midazolam and Remifentanil During Arteriovenous Fistula Placement Procedure and Monitored Anesthesia Care
Brief Title: The Use of Midazolam and Remifentanil During Dialysis Access Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Collaborators: Trakya University (Other)
Responsible Party: Principal Investigator, Ayse Baysal, Associate Professor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013.1/28(#)
Record Dates: First submitted 2019-11-28; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Sedative Adverse Reaction; Analgesic Adverse Reaction; Midazolam Adverse Reaction; Adverse Reaction to Drug; Patient Satisfaction; Chronic Kidney Diseases; Arteriovenous Fistula
Keywords: Midazolam; Remifentanil; Benzodiazepine; Opioid; Chronic Kidney Diseases; Analgesia; Sedation; Adverse Reaction; Patient Satisfaction; Arteriovenous Fistula
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Patient Satisfaction; Renal Insufficiency, Chronic; Arteriovenous Fistula; Agnosia | interventions — Midazolam; Remifentanil

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized clinical study. The patients were divided into two groups with a 1: 1 allocation and sealed envelope randomization method. Both groups of patients received intravenous midazolam, in Group 1, intravenous midazolam was administered continuously whereas, in Group 2, intravenous midazolam was administered as intermittent bolus doses. Both groups received intravenous remifentanil bolus doses as a rescue medication.
Who Masked: Participant, Care Provider
Masking Description: This study was a single-blinded controlled study because the sedation and analgesia were administered by anesthesiology residents who were unaware of the technique and the study protocol, however, the protocol was known by the experienced anesthesiologist who was attending the case and collecting the data during the procedure. The preparation of midazolam and remifentanil solutions and installation of the infusion devices were done by an anesthesiologist who was blinded for the study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): In Group 1(n=50); continuous infusion of intravenous midazolam (Dormicum, Deva Pharmaceutical, Turkey) at a dose of 0.02 to 0.04 mg/kg/h was started at the beginning of the operation and the dose was adjusted depending on pain level and sedation level using appropriate scales for monitoring throughout the surgical time period. An intravenous bolus dose of midazolam at a dose of 0.015 mg/kg was administered before the start of the surgery. A rescue medication of intravenous bolus dose of remifentanil at a concentration of 5 μg/mL was used every 5 to 10 minutes in doses of 1 to 3 mL if necessary for pain scores greater than 3. The medications were stopped prior to the end of the surgery.
  Interventions: Drug: Midazolam intravenous injection; Drug: Remifentanil intravenous bolus dose
- Group 2 (Active Comparator): in Group 2 (n=49), intravenous bolus doses of midazolam at a dose of 0.015 mg/kg every 10 minutes were administered at the beginning of the operation and the dose was adjusted depending on pain level and sedation level using appropriate scales for monitoring throughout the surgical time period. An intravenous bolus dose of midazolam at a dose of 0.015 mg/kg was administered before the start of the surgery. A rescue medication of intravenous bolus dose of remifentanil at a concentration of 5 μg/mL was used every 5 to 10 minutes in doses of 1 to 3 mL if necessary for pain scores greater than 3. The medications were stopped prior to the end of the surgery.
  Interventions: Drug: Midazolam intravenous injection; Drug: Remifentanil intravenous bolus dose

INTERVENTIONS:
Drug: Midazolam intravenous injection — The midazolam was prepared as 5 mg midazolam in 20 mL syringe of 5% dextrose water solution (0.25 mg/mL) in both arms. Both groups of patients received an intravenous bolus dose of midazolam was administered before the start of the surgery. In Group 1, continuous infusion of intravenous midazolam was started and in Group 2, intravenous bolus doses of midazolam were administered. The doses were adjusted depending on pain level and sedation level using appropriate scales for monitoring during the surgical time period. The drip rate was adjusted according to pain intensity. The infusion of drugs was discontinued at the end of the procedure.
  Other Names: Dormicum, Deva Pharmaceutical, Turkey
Drug: Remifentanil intravenous bolus dose — A remifentanil infusion was prepared as follows; 0.5 mg remifentanil was added into 100 mL of 0.9% saline at a concentration of 5 μg/mL. The preparation of remifentanil solution and installation of the device was done by an anesthesiologist who was blinded for the study groups. The dose and number of patients that required remifentanil were recorded. The infusion of drugs was discontinued at the end of the procedure. A rescue medication of intravenous remifentanil bolus dose was used as 1 to 3 mL (5 μg or 15 μg) every 5 minutes if necessary for pain scores greater than 3. This infusion was prepared prior to the use during the study and was discontinued at the end of the procedure.
  Other Names: Ultiva, Glaxo Smith Kline Pharmaceutical, England

SUMMARY:
BACKGROUND: Sedation and analgesia are related to unexpected adverse events in chronic renal failure patients undergoing arteriovenous fistula placement procedures under monitored anesthesia care (MAC).

OBJECTIVE: Our goal was to investigate and compare the sedation and analgesia related effects and adverse effects of continuous intravenous use of midazolam and intermittent bolus doses of midazolam while intravenous remifentanil is used as a rescue medication in patients with chronic renal failure.

DETAILED DESCRIPTION:
BACKGROUND: Sedation and analgesia are related to unexpected adverse events in chronic renal failure patients undergoing arteriovenous fistula placement procedures under monitored anesthesia care (MAC).

OBJECTIVE: Our goal was to investigate and compare the sedation and analgesia related effects and adverse effects of continuous intravenous use of midazolam to intermittent bolus doses of midazolam while intravenous remifentanil is used as a rescue medication in patients with chronic renal failure.

DESIGN: From a total of 116 patients, 99 patients with chronic renal failure undergoing arteriovenous fistula procedures were included in a prospective randomized study.

SETTINGS: Two tertiary care hospitals. PATIENTS: The patients were divided into Group 1 (continuous)(n=50); patients receiving intravenous midazolam infusion at a dose of 0.02 to 0.04 mg/kg/h and Group 2 (intermittent)(n=49); patients receiving intermittent intravenous bolus doses of 0.015 mg/kg every 10 minutes.

MAIN OUTCOME MEASURES: Primary outcomes were; 1- The total amount of doses of the use of midazolam and remifentanil in both groups of patients, 2- The evaluation of satisfaction of patient and surgeon at the end of the operation, in the recovery room during the period of recovery from sedation and before discharge. Other outcome measures include; the sedative, analgesic and hemodynamical effects of sedative medications that were compared in both groups of patients during the operation time period. The hospital stay duration was recorded and compared between groups. The maximum dose of midazolam was limited to 4 mg intravenously. The intensity of pain was assessed using a verbal numerical sedation scale (range 1 to 10) (VNRS) and the sedation level was recorded by Modified Observer's Assessment of Alertness/Sedation Scale (MOSS/A) (range 0 to 6). MOSS/A Scale includes; Score 0: Does not respond to deep stimulus, Score 1: Does not respond to mild prodding or shaking, Score 2: Responds only after mild prodding or shaking, Score 3: Responds only after name is called loudly and/or repeatedly, Score 4: Lethargic response to name spoken in normal tone, Score 5: Responds readily to name spoken in normal tone, Score 6: Agitated. An intravenous bolus dose of remifentanil as a rescue medication was administered for pain scores greater than 3 at a dose of 5µg/mL. Adverse events were recorded. Patient satisfaction level depending on the experience in general were evaluated at discharge from 0 to 4 point numerical scale: 0 = extremely dissatisfied; 1 = dissatisfied; 2 = neither satisfied nor dissatisfied; 3 = satisfied; 4 = extremely satisfied. Surgeon satisfaction level depending on the experience in general were evaluated at discharge from five-point numerical scale: 0 = extremely poor; 1 = poor; 2 = fair; 3 = good; 4 = excellent.

SAMPLE SIZE: The sample size was calculated based on a power of 80% and a 5% type-I error and for each group, thirty patients were required.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Forty-three to eighty-one years of age,
2. ASA status: American Society of Anesthesiologist (ASA) status I-III,
3. The diagnosis: A diagnosis of chronic renal failure,
4. The operation type: An arteriovenous fistula procedure

Exclusion Criteria:

1. Body mass index greater than 40 that are considered morbidly obese patients,
2. Lung disorders leading to severe respiratory insufficiency such as; severe asthma, chronic obstructive lung disease,
3. Severe cardiovascular insufficiency or dysfunction,
4. Insulin-dependent diabetes mellitus,
5. Severe hepatic diseases,
6. ASA status of 4 and 5,
7. Neurologic disorders such as; the presence of epilepsy, arterial aneurysm, intracranial mass,
8. Patients complaining about intense pain before the procedure and patients with a history of long term opioid use or chronic pain,
9. Patients with a history of allergy to the study drugs,
10. Patients without written informed consent.

Ages: 43 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-08-28 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
The amount of total use of midazolam and remifentanil drug consumptions in milligrams during operation time period. | Through the operative time period up to two hours of time.
  The comparison of total use of midazolam and remifentanil drug consumptions in milligrams during operation time period between the two groups.
The evaluation of satisfaction of patient and surgeon by a questionnaire at the end of operation. | The collection of questionnaire at the end of operation in recovery room after recovery from sedation in a total of ten minutes time.
  The evaluation and comparison of satisfaction of patient and surgeon at the end of operation by a questionnaire between the two groups. Patient satisfaction level depending on the experience in general was evaluated at discharge from 0 to 4 point numerical scale: 0 = extremely dissatisfied; 1 = dissatisfied; 2 = neither satisfied nor dissatisfied; 3 = satisfied; 4 = extremely satisfied. Surgeon satisfaction level depending on the experience in general was evaluated at discharge from five point numerical scale: 0 = extremely poor; 1 = poor; 2 = fair; 3 = good; 4 = excellent.
Modified Observer's Assessment of Alertness/Sedation Scale (MOSS/A) Scale | Through the operative time period up to two hours of time.
  The comparison of level of sedation using MOSS/A scale that ranges from 0 to 6, with a score of 6 defined as awake or minimally sedated, and a score of 0 defined as general anesthesia every 10 to 15 minutes between the two groups.
Modified Observer's Assessment of Alertness/Sedation Scale (MOSS/A) Scale | Through the operative time period up to two hours of time.
  Repeated measure analysis of level of sedation by the use of the collected MOSS/A scale that ranges from 0 to 6, with a score of 6 defined as awake or minimally sedated, and a score of 0 defined as general anesthesia every 10 to 15 minutes within groups.
Verbal Numerical Rating Scale | Through the operative time period up to two hours of time.
  The comparison of level of pain using Verbal Numerical Rating Scale (VNRS; 0= no pain, 10=the worst possible pain imaginable) scale every 10 to 15 minutes between the two groups.
Verbal Numerical Rating Scale | Through the operative time period up to two hours of time.
  Repeated measure analysis of level of sedation by the use of the collected Verbal Numerical Rating Scale (VNRS; 0= no pain, 10=the worst possible pain imaginable) scale every 10 to 15 minutes between the two groups.
Recovery time | Through the recovery room time period before discharge up to one hour time.
  The comparison of recovery time duration presented in minutes unit of time between the two groups.
Hospital stay | Through the duration of stay in hospital before discharge up to seventy two hours time.
  The comparison of hospital stay duration presented in hours unit of time between the two groups.
Systolic blood pressure values during operation and in the recovery room. | Through the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time.
  The comparison of systolic blood pressure in mmHg unit values every 15 minutes between the two groups.
Heart rate values during operation and in the recovery room. | Through the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time.
  The comparison of heart rate values in beats per minute unit every fifteen minutes between the two groups.
Pulse oximetry values during operation and in the recovery room. | Through the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time.
  The comparison of pulse oximetry values in percent unit every fifteen minutes between the two groups.
Adverse events during operation and in the recovery room. | Through the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time.
  Number of Participants With Adverse Events as Assessed by CTCAE Version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Gonul Sagiroglu, MD, Study Director — Trakya University

IPD SHARING:
Plan to Share IPD: Yes
This is a prospective, randomized clinical study. Both groups of patients received intravenous midazolam in two different methods. The groups were assigned depending on the use of intravenous midazolam as a continuous infusion or intermittent bolus doses. In both groups, as a rescue medication, intravenous bolus doses of remifentanil was used. The titration of the doses of midazolam and remifentanil was done according to the use of pain intensity level and the sedation level evaluations. The primary outcome was the comparison of the total amount of doses of the use of midazolam and remifentanil in milligrams in both groups of patients and the comparison of the satisfaction of patients and surgeons using an appropriate questionnaire. The pain intensity and sedation level, hemodynamical effects, as well as adverse events, were compared in both groups of patients. The recovery time and hospital stay duration were compared between the two groups of patients.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available after registration and will be available upon request from the Clinical Study Director at any time after registration.
Access Criteria: Study Protocol and Statistical Package for the Social Sciences computer program data.

REFERENCES:
- [Background] Cole NM, Vlassakov K, Brovman EY, Heydarpour M, Urman RD. Regional Anesthesia for Arteriovenous Fistula Surgery May Reduce Hospital Length of Stay and Reoperation Rates. Vasc Endovascular Surg. 2018 Aug;52(6):418-426. doi: 10.1177/1538574418772451. Epub 2018 Apr 29. PMID 29706126
- [Background] Sa Rego MM, Inagaki Y, White PF. Remifentanil administration during monitored anesthesia care: are intermittent boluses an effective alternative to a continuous infusion? Anesth Analg. 1999 Mar;88(3):518-22. doi: 10.1097/00000539-199903000-00009. PMID 10071997
- [Background] Sun GQ, Gao BF, Li GJ, Lei YL, Li J. Application of remifentanil for conscious sedation and analgesia in short-term ERCP and EST surgery. Medicine (Baltimore). 2017 Apr;96(16):e6567. doi: 10.1097/MD.0000000000006567. PMID 28422846
- [Background] Wyne A, Rai R, Cuerden M, Clark WF, Suri RS. Opioid and benzodiazepine use in end-stage renal disease: a systematic review. Clin J Am Soc Nephrol. 2011 Feb;6(2):326-33. doi: 10.2215/CJN.04770610. Epub 2010 Nov 11. PMID 21071517
- [Background] Ahuja V, Mitra S, Kazal S, Huria A. Comparison of analgesic efficacy of flupirtine maleate and ibuprofen in gynaecological ambulatory surgeries: A randomized controlled trial. Indian J Anaesth. 2015 Jul;59(7):411-5. doi: 10.4103/0019-5049.160937. PMID 26257413
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- [Result] Boonstra AM, Stewart RE, Koke AJ, Oosterwijk RF, Swaan JL, Schreurs KM, Schiphorst Preuper HR. Cut-Off Points for Mild, Moderate, and Severe Pain on the Numeric Rating Scale for Pain in Patients with Chronic Musculoskeletal Pain: Variability and Influence of Sex and Catastrophizing. Front Psychol. 2016 Sep 30;7:1466. doi: 10.3389/fpsyg.2016.01466. eCollection 2016. PMID 27746750
- [Result] Beathard GA, Urbanes A, Litchfield T, Weinstein A. The risk of sedation/analgesia in hemodialysis patients undergoing interventional procedures. Semin Dial. 2011 Jan-Feb;24(1):97-103. doi: 10.1111/j.1525-139X.2011.00844.x. PMID 21338400
- [Result] Son A, Mannoia K, Herrera A, Chizari M, Hagdoost M, Molkara A. Dialysis Access Surgery: Does Anesthesia Type Affect Maturation and Complication Rates? Ann Vasc Surg. 2016 May;33:116-9. doi: 10.1016/j.avsg.2015.12.005. Epub 2016 Mar 8. PMID 26965819
- [Result] Niscola P, Scaramucci L, Vischini G, Giovannini M, Ferrannini M, Massa P, Tatangelo P, Galletti M, Palumbo R. The use of major analgesics in patients with renal dysfunction. Curr Drug Targets. 2010 Jun;11(6):752-8. doi: 10.2174/138945010791170879. PMID 20041843
- [Result] Hatzidakis AA, Charonitakis E, Athanasiou A, Tsetis D, Chlouverakis G, Papamastorakis G, Roussopoulou G, Gourtsoyiannis NC. Sedations and analgesia in patients undergoing percutaneous transhepatic biliary drainage. Clin Radiol. 2003 Feb;58(2):121-7. doi: 10.1053/crad.2002.1128. PMID 12623040
- [Result] Coyle TT, Helfrick JF, Gonzalez ML, Andresen RV, Perrott DH. Office-based ambulatory anesthesia: Factors that influence patient satisfaction or dissatisfaction with deep sedation/general anesthesia. J Oral Maxillofac Surg. 2005 Feb;63(2):163-72. doi: 10.1016/j.joms.2004.10.003. PMID 15690283